CLINICAL TRIAL: NCT06681987
Title: Simulation in Preeclampsia and Eclampsia Management: Innovative Approaches in Midwifery Education
Brief Title: Innovative Approaches in Midwifery Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Lecturer, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-95531838-050.99-116027
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Simulation Training
Keywords: pre-eclampsia; simulation; midwifery
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- simulation (Experimental): One group of students will practice computer-based simulation for pre-eclampsia and eclampsia case management skills using a high-fidelity simulator (n = 15) (subgroups n=3), while the other group will practice with a low-fidelity model (n = 15; subgroups n=3). In the first stage, the case will be written for the high-fidelity simulator and will be submitted to the opinions of experts in the field. After the necessary arrangements are made, the groups will be randomized and allocated. In the second stage, the experimental group will be presented with a virtual reality simulator, and the control group will be presented with a case example of preeclampsia and eclampsia with a low-level simulator. In order to evaluate and increase the teamwork skills of the students in the experimental and control groups, the students will be divided into subgroups of three.
  Interventions: Behavioral: simulation training
- control (No Intervention): application will be made in a low reality model

INTERVENTIONS:
Behavioral: simulation training — One group of students will practice computer-based simulation for pre-eclampsia and eclampsia case management skills using a high-fidelity simulator (n = 15) (subgroups n=3), while the other group will practice with a low-fidelity model (n = 15; subgroups n=3). In the first stage, the case will be written for the high-fidelity simulator and will be submitted to the opinions of experts in the field. After the necessary arrangements are made, the groups will be randomized and allocated. In the second stage, the experimental group will be presented with a virtual reality simulator, and the control group will be presented with a case example of preeclampsia and eclampsia with a low-level simulator. In order to evaluate and increase the teamwork skills of the students in the experimental and control groups, the students will be divided into subgroups of three.
  Arms: simulation

SUMMARY:
In midwifery education, simulations often cover areas such as labor and neonatal care, emergency management, birth complications, and routine maternal care. High-reality simulation mannequins allow students to practice a variety of skills, such as managing normal deliveries and complications, providing care during caesarean section, or performing initial interventions on the newborn. It increases knowledge, critical thinking, confidence and competence, especially in obstetric emergencies where clinical exposure may be limited. Simulation supports the development of both technical and non-technical skills, including teamwork. To be effective, simulation needs to include briefing (feedback), good communication, observation, repetition, reflection and evaluation. However, it remains a valuable tool for creating safe learning environments that mimic real clinical scenarios without patient risk. It helps students practice staying calm and working in an organized manner in the face of stressful situations they may encounter in real life.

DETAILED DESCRIPTION:
Instead of the tension and pressure that can be experienced in real patient care, simulations alleviate students' fear of making mistakes by providing a safe environment. This reduces stress and allows students to feel more relaxed. As students have the opportunity to learn from their mistakes and make amends, they can act more confidently when faced with stressful situations. However, it should not be ignored that simulation may cause stress in some students. Since simulations confront students with situations that are close to real clinical scenarios, they may cause students to feel intense pressure, especially in complex or emergency situations. Although there are no real patients in the simulation environment, the realism of the scenarios and the evaluation of their performance by the instructors may increase the stress level in some students. However, this type of stress is usually considered as part of a positive learning process because it allows students to experience less stress when they face similar situations later on. Managing stress during simulation training is also an important part of the training. Post-simulation feedback and evaluation sessions help students to review their emotional and psychological state. This process can help students to evaluate themselves, develop strategies to cope with stress and feel less anxious in the future. In addition, teamwork and collaboration among students during the simulation can also be effective in stress management. Their ability to communicate within the team, receive support and solve problems together contributes to students' relaxation by reducing stress levels.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the research
* To have successfully passed all courses
* The student does not have visual and hearing impairment problems
* Studying in the 7th academic semester

Exclusion Criteria:

* Refusing to participate in the research
* Incomplete/incorrect completion of data collection tools
* Receiving a psychiatric diagnosis such as anxiety disorder
* Excessive stress
* Problems with hand-eye coordination

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — midwifery students are girls.
Enrollment: 30 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Problem Solving skills | one day after the training
  Problem solving skill scores will increase after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Ibrahim Çeçen University Faculty of Health Sciences, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It may not be appropriate to share data in order to protect participants' privacy and fulfill ethical obligations. As participants do not know that their data will be shared with others, this may violate their privacy.

REFERENCES:
- [Background] Pajohideh ZS, Mohammadi S, Keshmiri F, Jahangirimehr A, Honarmandpour A. The effects of normal vaginal birth simulation training on the clinical skills of midwifery students: a quasi-experiment study. BMC Med Educ. 2023 May 19;23(1):353. doi: 10.1186/s12909-023-04319-9. PMID 37208680